| | CLINICAL RESEARCH TEMPIATE | Document No: | Page 1/12 |
|---|---|---|---|
| | | CR-TMP-01.22 | Version: 1.0 |
| Title: | | | |
| Clinical Research: Statistical Ana | atistical Analysis Plan Template | | |

Unique Protocol ID: NOWDx COVID-19 Antibody POC

H

NOWDx Test for the Detection of Antibodies to COVID-19

**Brief Title:** 

NCT Number: NCT04690413

Document Date: September 01, 2020

**⊗** N○Wdiagnostics

CLINICAL RESEARCH TEMPLATE

Document No:

Version: 1.0 Page 1/12

Clinical Research: Statistical Analysis Plan Template

## Statistical Analysis Plan

Project Name
NOWDx COVID-19 EUA Blood Test CLIA Waiver Trial; IRB # Pro00045452

Project Personnel
Sponsor Principal Investigator: Beth Cobb
Person(s) performing statistical analyses: Beth Cobb, Shincy Koodathil, Kelsi Thurman, Jessica Thomas, Lexie Hopper

| Study Design | sign | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Cohort<br># | Cohort Cohort Name | Cohort<br>Size | Prospective or<br>Retrospective? | Case or<br>Control? | Inclusion<br>Criteria | Exclusion<br>Criteria | Data to be collected | Sub- |
| ~ | Persons who have tested positive for COVID-19 with an emergency use authorized molecular (PCR) test and can furnish said test report; ≥ 7 days post emergency use authorized molecular (PCR) test | 30 | Prospective | Case | Persons who have tested positive for COVID-19 with an emergenc y use authorized molecular (PCR) test and can furnish said test report; ≥ 7 days post | Persons <18 years old; persons with limited or no reading skills; persons who previously participated in a NOWDx study; < 7 days post emergency use authorized molecular (PCR) test | Phone Screening Script Responses; Screening/Enrolm ent Log; ICFs; Surveys; CRFs; Study Visit Checklist and Incentive Receipt forms; EUA molecular (PCR) test report; AE/SAE forms | N/A |

| <b>NOWdiagnostics</b> |
|-----------------------|
| <b>5</b> |

Document No:


Version: 1.0

Clinical Research: Statistical Analysis Plan Template Title:

| | N/A |
|---|---|
| | Phone Screening<br>Script Responses;<br>Screening/Enrolm<br>ent Log; ICFs;<br>Surveys; CRFs;<br>Study Visit<br>Checklist and<br>Incentive Receipt<br>forms; EUA<br>molecular (PCR)<br>test report;<br>AE/SAE forms |
| | Persons <18 years old; persons with limited or no reading skills; persons who previously participated in a NOWDx study; > 6 days post emergency use authorized molecular (PCR) test |
| emergenc<br>y use<br>authorized<br>molecular<br>(PCR) test | Persons who have tested positive for COVID-19 with an emergenc y use authorized molecular (PCR) test and can furnish said test report; 0-6 days post emergenc y use authorized |
| | Case |
| | Prospective |
| | 30 |
| | Persons who have tested negative for COVID-19 with an emergency use authorized molecular (PCR) test and can furnish said test report; 0-6 days post EUA molecular (PCR) test |
| | 8 |

The contents of this document are **CONFIDENTIAL** and **PROPRIETARY** to Now Diagnostics, Inc. and shall not be disclosed, disseminated, copied, and used except for purposes expressly authorized in writing by Now Diagnostics, Inc.

| Ń |
|---|
| .2 |
| to |
| Ö |
| Ē |
| 0 |
| O |
| - |
| > |
| $\leq$ |
| 7 |
| 4 |
| THE STATE OF THE S |

Title:

CLINICAL RESEARCH TEMPLATE


Document No:


Clinical Research: Statistical Analysis Plan Template

| Samples<br>Reporting | Samples to be Collected (Note: must include the 'complete spectrum of patient characteristics' – see FDA Statistical Guidance on Reporting Results from Studies Evaluating Diagnostic Tests) | e: must include<br>es Evaluating D | the 'complete<br>Diagnostic Tes | spectrum of , sts) | patient characteristi | cs' – see FDA Stati | istical Guidance on |
|---|---|---|---|---|---|---|---|
| Cohort<br># | Cohort Name | Type(s) of<br>Specimens | Tube<br>type(s) | Quantity | Collection<br>Procedure | Storage<br>Procedure | Handling<br>Procedure |
| ~ | Persons who have tested positive for COVID-19 with an emergency use authorized molecular (PCR) test and can furnish said test report; ≥ 7 days post emergency use authorized molecular (PCR) test | Blood; plasma | EDTA | 1 EDTA | Standard<br>phlebotomy;<br>fingerstick | ≥ -20°C | Study sites will ship plasma from EDTA tubes to NOWDx |

| | CI INICAL BESEABCH TEMBI ATE | Document No: | Page 4/12 |
|---|---|---|---|
| Title: | | | |
| Clinical Research: Statistical Ana | nalysis Plan Template | | |

| Reference Standard Method: N/A Non-Reference Standard/Comparative Method: N/A Power/Sample size calculations: Sample size is determined by FDA EUA Guidance for serology assays. Intended Use Sites (minimum = 3) Study Site Address Study Site |
|---|

The contents of this document are **CONFIDENTIAL** and **PROPRIETARY** to Now Diagnostics, Inc. and shall not be disclosed, disseminated, copied, and used except for purposes expressly authorized in writing by Now Diagnostics, Inc.

| | S |
|---|-----|
| | JOS |
| | age |
| • | 2 |

Document No: Page 5/12


Title:

Clinical Research: Statistical Analysis Plan Template

| Clinical Research<br>Solutions, LLC | 2075 Pleasant Plains<br>Extension, Jackson, TN<br>38305 | PI: Melanie Hoppers, M.D.<br>Site operators 1& 2: Aubrey Walgren; William Edwards;<br>Hannah Wells | I.D.<br>brey Walgren; Wil | lliam Edwar | ds; Both | |
|---|---|---|---|---|---|---|
| | Ph. 731-984-8400 | | | | | |
| Comprehensive<br>Clinical<br>Research, LLC | 603 Village Blvd. Suite<br>301. West Palm Beach,<br>FL 33409 (561) 478-<br>3177; (561) 683-1331<br>(24 hours) | PI: Ronald Ackerman, MD, FACOG<br>Site operators 1& 2: Diana Mann; Tomeko Heard | MD, FACOG<br>ana Mann; Tomek | o Heard | Both | |
| Del Sol Research<br>Management,<br>LLC | 5700 East Pima Street,<br>Suite A. Tucson, AZ<br>85712<br>Ph. 520-257-3881 | PI: Carl F. Diener, MD<br>Site operators 1 & 2: Antonia Garcia; Krissa Goodin | ntonia Garcia; Kris | ssa Goodin | Both | |
| NOWDx Test/Devic | NOWDx Test/Device – ADEXUSDx® COVID-19 Test | 9 Test | | | _ | |
| Intended Use | | | Intended<br>Operator<br>Experience | Test<br>Setting | Controls<br>Applied? | Specimen<br>Acceptance<br>Criteria |
| The ADEXUSDx® immunoassay inter SARS-CoV-2 in ht ADEXUSDx® COV identifying individua | The ADEXUSDx® COVID-19 Test is an <i>in vitro</i> lateral flow immunoassay intended for qualitative detection of total antibodies to SARS-CoV-2 in human whole blood(venous and fingerstick). The ADEXUSDx® COVID-19 Test is intended for use as an aid in identifying individuals with an adaptive immune response to SARS- | an in vitro lateral flow tion of total antibodies to us and fingerstick). The for use as an aid in une response to SARS- | CLIA Waived<br>operator | Point of<br>Care | Internal and External Controls (applied once | Capillary blood/<br>venous whole blood<br>volume sufficient to<br>fill the Fill Zone and<br>reach the Fill Line |

| <b>M</b> ON <b>Q</b> | agnostics |
|----------------------|-----------|
| <b>S</b> | |
| 0 | O<br>Z |
| | D |

Document No:

Version: 1.0 Page 6/12

Title: Clinical Research: Statistical Analysis Plan Template

| CoV-2, indicating recent or prior infection. for how long antibodies persist following informantibodies confers protective immunity. whole blood (EDTA) and fingerstick specin patient care settings authorized to perform | CoV-2, indicating recent or prior infection. At this time, it is unknown for how long antibodies persist following infection and if the presence of antibodies confers protective immunity. Testing of human venous whole blood (EDTA) and fingerstick specimens can be conducted in patient care settings authorized to perform CLIA waived tests. | At this time, it is unknown ection and if the presence Testing of human venous nens can be conducted in CLIA waived tests. | | for each lot of tests) |
|---|---|---|---|---|
| Reference Standard Test/Device | est/Device | | | |
| Intended Use | Intended Operator Experience | Test Setting | Controls Applied? | Specimen Acceptance Criteria |
| N/A | N/A | N/A | N/A | N/A |
| Non-Reference Stand | <br> Non-Reference Standard/Comparative Method Test/Device | d Test/Device - N/A | | |
| Intended Use | Intended Operator Texperience | Test Setting | Controls Applied? | Specimen Acceptance Criteria |
| N/A | | N/A | N/A | N/A |
| FLEX Studies (to ident<br>Waiver Guidance 2020 | tify potential device deficie | encies, including failur | es and determine the r | FLEX Studies (to identify potential device deficiencies, including failures and determine the robustness of the test system; See 6-8, CLIA Waiver Guidance 2020 |
| Operator error FLEX studies | studies | Specimen volume | Specimen volume, reading time; unique test characteristics | test characteristics |
| Specimen integrity and | Specimen integrity and handling FLEX studies | N/A | | |
| Reagent Integrity/Visibility FLEX studies | oility FLEX studies | N/A | | |

| diagnostics |
|-------------|
| NON |

Document No: Page

Page 7/12 Version: 1.0

Title:

Clinical Research: Statistical Analysis Plan Template

| Hardware, software and electronics integrity FLEX studies | N/A |
|---|---|
| Stability of calibration and internal controls FLEX N/A studies | N/A |
| Environmental factors FLEX studies | Temperature and Humidity; Light |
| Other | N/A |
| Cross-Reactivity | |

Not required due to performance of the test in the internal validation study; submitted to FDA on 05/29/2020

#### Interference

N/A

Method Comparison Studies (Min: 3 sites; 2 operators; equal distribution b/w operators (min: 10 pos, 10 neg each operator); 30 positive samples, 30 negative samples); PERFORM site specific and overall analyses; also PERFORM for fingerstick and venous sample results separately in comparison to comparator, not to each other) The results from this study should be presented as sensitivity and specificity as compared to the comparator method and should have a PPA of 90% and NPA of 95%; 2x2 table format; data to be stratified by days since PCR result; data to be presented separately for each matrix testing method (fingerstick and venous whole blood).

professional operators); include samples of all concentrations; 60 weak positive aliquots and 60 weak negative aliquots evenly distributed p.29); Goal: find concentrations where the indicator (colored line) is observed 95% (weak positive) or 5% (weak negative) of the time by Determining Device Performance with Analyte Concentrations Near the Cutoff (Dilution studies (see 2020 CLIA Waiver guidance across 3 sites; MASKED & order randomized TO professional OPERATORS)

N/A

### Reproducibility Studies

₹ Z



Document No:


Clinical Research: Statistical Analysis Plan Template

# Interim Analyses (See CR-WI-01.21: Clinical Research: Statistical Analysis Plan)

A bi-weekly interim analysis will be performed, and a presentation will be sent to the CEO of an overview of study recruitment to date. At the discretion of the Director of Operations, said presentations may also include study recruitment per cohort per site, sensitivity & specificity data, and any updates regarding preparation for EUA submission.

Purpose of interim analyses: to monitor completion rate of studies and test performance

Decisions to be made as a result of interim analyses: increase study sites, interim study visit monitoring, retraining, etc.

#### Derived variables

#### Software

We will use Microsoft Office 365 Excel (Version 16.0 or latest version) to perform statistical analyses of data.

### Data Summarization

Demographic and clinical characteristics of cohorts will be summarized (in text or table form). Demographic data to be summarized may include gender diversity, ethnicity and racial diversity, age diversity, and education diversity.

# Ethnicity and Racial Diversity (RECORD FOR EACH STUDY SITE & COLLECTIVELY):

| | | | | | Ethnic | Ethnic Categories | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Not H | Not Hispanic or Latir | . Latino | His | Hispanic or Latino | atino | | Jnknown/Not Reported Ethnicity | d Ethnicity | Total |
| Racial<br>Categories | Female | Male | Unknown<br>/Not<br>Reported | Female | Male | Unknown<br>/Not<br>Reported | Female | Male | Unknown<br>/Not<br>Reported | |
| White | | | | | | | | | | |

| S |
|------|
| Stic |
| 2 |
| 0 |
| 0 |
| Z |
| 0 |

Document No:


Clinical Research: Statistical Analysis Plan Template Title:

| Black or<br>African<br>American | American<br>Indian/Alaska<br>Native | Asian | Native<br>Hawaiian or<br>Other Pacific<br>Islander | Unknown | Total |
|---|---|---|---|---|---|

Age Diversity (RECORD FOR EACH STUDY SITE & COLLECTIVELY):

| Age Range (in years) | # of Males | # of Females |
|----------------------|------------|--------------|
| 18-24 | | |
| 25-34 | | |
| 35-44 | | |
| 45-54 | | |
| 55-64 | | |

| NOWdiagnostics | CLINICAL RESEARCH TEMPLATE | Document No: |
|----------------|----------------------------|--------------|
| Title: | | |

Clinical Research: Statistical Analysis Plan Template

**65**+


Education Diversity (RECORD FOR EACH STUDY SITE & COLLECTIVELY):

| | _ | _ | | | | | | | | _ |
|---|---|---|---|---|---|---|---|---|---|---|
| # of Females | | | | | | | | | | |
| # of Males | | | | | | | | | | |
| Highest degree/level of school completed # of Ma | No schooling completed | Some grade school, no diploma | High school graduate, diploma, or the equivalent (for example: GED) | Some college credit, no degree | Trade/technical/vocational training | Associate degree | Bachelor's degree | Master's degree | Doctorate degree | |

| | | Positive | Negative |
|---------------------|----------|----------|----------|
| | Positive | А | Q |
| NOWDX COVID-19 lest | Negative | C | В |

Comparator Test

Sensitivity (AKA the true positive rate): A/(A+C) Specificity (AKA the true negative rate): B/(B+D)

NOWdiagnostics

Title:

CLINICAL RESEARCH TEMPLATE

Document No: CR-TMP-01.22


Clinical Research: Statistical Analysis Plan Template

| | | ຮື | Candidate Device Results | |
|---|---|---|---|---|
| Days since EUA PCR<br>Test | Number of Samples<br>Tested | Total Antibody Positive<br>Results | Total Antibody PPA | 95% CI |
| | 4 | В | a/A (%) | |
| | Ω | q | b/B (%) | |
| 14-20 days | ပ | O | c/C (%) | |
| | ٥ | σ | d/D(%) | |

SAP Amendment Process (See CR-WI-01.21: Clinical Research: Statistical Analysis Plan)

The SAP and any subsequent revisions must be version controlled and recorded in the SAP Revision History Table. The SAP Revision History Table records the following information:

- Author of change
  - Version number
    - Version date

The final SAP version must be approved by all named approvers. Section/content changed

#### SAP Training

work. Personnel should pose questions to PI to clarify any misunderstandings or areas of confusion. Training should be documented using All project personnel will review the SAP and all associated procedures or project documents in detail prior to performance of any project the Statistical Analysis Plan Training Log CR-LOG-01.25.

| | CIINICAI BESEABCH TEMBIATE | Document No: | Page 12/12 |
|----------------|----------------------------|--------------|--------------|
| A VACING SILCS | | | Version: 1.0 |
| itle: | | | |

Author of this Statistical Analysis Plan (Name) and, if different to that of the Sponsor Principal Investigator, their telephone & email contact details
Shincy Koodathil; 479-966-4514; Shincy Koodathil@nowdx.com

Clinical Research: Statistical Analysis Plan Template

Approved by:

| | $\widehat{\mathbf{L}}$ |
|---|------------------------|
| | /estigator (F |
| | ≧ |
| | Principal |
| • | Sponsor |

| 09/01/3000 | Date |
|-------------|------|
| ask of cobb | Name |

Director of Operations (if different than Sponsor PI)

Date

Name